CLINICAL TRIAL: NCT00428012
Title: Quality of Life Therapy for Adults With ESRD Awaiting Renal Transplantation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Rodrigue, Associate Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R21 DK77322 (completed); R21DK077322 (NIH)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: End-stage Renal Disease
Keywords: quality of life, kidney transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- QOLT (Experimental): Quality of Life Therapy (QOLT) 8 weekly individual counseling sessions
  Interventions: Behavioral: Quality of Life Therapy
- ST (Active Comparator): Supportive Therapy (ST) 8 weekly individual counseling sessions
  Interventions: Behavioral: Supportive Therapy
- Standard Care (No Intervention)

INTERVENTIONS:
Behavioral: Quality of Life Therapy — 8 weekly individual counseling sessions
  Arms: QOLT
Behavioral: Supportive Therapy — 8 weekly individual counseling sessions
  Arms: ST

SUMMARY:
The purpose of this study is to determine whether psychological intervention is effective in improving quality of life, mood, and relationships among adults with end-stage renal disease who are awaiting kidney transplantation.

DETAILED DESCRIPTION:
Despite known quality of life (QOL) deficits associated with end-stage renal disease (ESRD), there have been very few attempts to develop strategies to improve QOL in adults with ESRD awaiting renal transplantation. The long-term goal of this research program is to better understand how QOL can be enhanced, to identify the mechanisms underlying QOL changes, to identify which patients benefit most from QOL intervention, and to determine whether QOL benefits can extend beyond transplantation. The objective of this research is to determine the effectiveness, feasibility and applicability of Quality of Life Therapy (QOLT) in treating adults with ESRD awaiting renal transplantation. In a recent small, single-center clinical trial, we demonstrated that QOLT can improve QOL, psychological functioning, and social intimacy in patients awaiting lung transplantation. We now seek to examine whether this intervention can be effectively adapted and implemented with adults with ESRD who are awaiting renal transplantation. The central hypothesis is that by targeting improvements in specific life domains, QOLT yields significant clinical benefits in QOL, psychological functioning, and the patient-caregiver relationship. This hypothesis is being tested by pursuing three specific aims: 1) Determine the effectiveness of QOLT; 2) Examine the differential effectiveness of QOLT by race (White, African American); and 3) Assess the feasibility of a multisite R01 application. Under the first aim, adults with ESRD awaiting renal transplantation are being randomized to receive QOLT, Supportive Therapy (ST), or Standard Care (SC). Primary outcomes are changes in QOL, psychological functioning, and social intimacy at 1 and 12 weeks post-treatment. Under the second aim, the relationship between race and intervention outcomes will be closely examined. Under the third aim, attrition rates, reasons for attrition, therapist adherence to treatment protocols, and participant satisfaction ratings are being gathered to assess the need for protocol changes prior to developing a larger, multisite clinical trial R01 application. This study is innovative because it is among the first to evaluate a theoretically-driven psychological intervention to specifically improve QOL in the context of ESRD and renal transplantation. The research is significant because it is expected to advance and expand understanding of how QOL can be improved in patients with ESRD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 21 and 70 years of age
* Diagnosis of ESRD
* Wait-listed for deceased donor renal transplantation (primary transplant only)
* White or African American race
* Signed informed consent
* Primary caregiver identified as spouse or domestic partner
* Resides within 60 minutes of transplant center

Exclusion Criteria:

* Prior recipient of renal transplantation
* Prior recipient of other solid organ transplantation
* Wait-listed for combined kidney-pancreas transplantation
* Current substance abuse or dependency
* Currently hospitalized
* Current recipient of psychological intervention services
* Mental retardation
* Substantial cognitive impairment (score of 23 or less on the Mini-Mental State Examination)
* Communication difficulties (speech, hearing) so substantial that they would prevent patient from participating actively in one of the interventions (determined by transplant social worker)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2007-01; Primary Completion 2009-07 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Primary: Scores on the following measures at 12 weeks post-intervention: Quality of Life Inventory, SF-36, KDQoL, CDC Activity Limitations Module, Hopkins Symptom Checklist, POMS, and Miller Social Intimacy Scale | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James R. Rodrigue, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- The Transplant Center, Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States